CLINICAL TRIAL: NCT03008109
Title: Short-term Injection of Recombinant Human Endostatin Plus EGFR-TKI as a Treatment of EGFR Mutation-positive Advanced Non-small Cell Lung Cancer
Brief Title: Endostar Plus EGFR-TKI（Epidermal Growth Factor Receptor-Tyrosine-Kinase Inhibitor） as a Treatment of EGFR Mutation-positive NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zaiwen Fan (Other Government)
Responsible Party: Sponsor-Investigator, Zaiwen Fan, Director of oncology department, Air Force General Hospital of the PLA
Organization: Air Force General Hospital of the PLA (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AirFGH
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Cancer; Lung Cancer, Nonsmall Cell
Keywords: EGFR-TKI; Recombinant human endostatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins

ARMS (1):
- EGFR-TK inhibitor plus RH-endostatin (Experimental): EGFR-TKI icotinib:125mg Tid RH-endostatin:15mg/m2 ,d1-7
  Interventions: Drug: EGFR-TK Inhibitor

INTERVENTIONS:
Drug: EGFR-TK Inhibitor
  Other Names: Recombinant human endostatin

SUMMARY:
EGFR Tyrosine-Kinase Inhibitor monotherapy is widely used in treatment of patients with EGFR mutation-positive Non-small cell lung cancer(NSCLC), In despite of the benefit of PFS （progression-free survival） , the OS （ overall survival） is limited extended. This study is aim to observe the safety and efficacy of the combination of an anti-angiogenic drug recombinant human-endostatin with EGFR TKI ,to find out a new strategy which may further extend the PFS and OS with a tolerated toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC,EGFR mutation positive,PS（performance status） 0-2,Patients were required to have one or more measurable lesions

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 18 month

REFERENCES:
- [Background] Gridelli C, Rossi A, Ciardiello F, De Marinis F, Crino L, Morabito A, Morgillo F, Montanino A, Daniele G, Piccirillo MC, Normanno N, Gallo C, Perrone F. BEVERLY: Rationale and Design of a Randomized Open-Label Phase III Trial Comparing Bevacizumab Plus Erlotinib Versus Erlotinib Alone as First-Line Treatment of Patients With EGFR-Mutated Advanced Nonsquamous Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2016 Sep;17(5):461-465. doi: 10.1016/j.cllc.2016.04.001. Epub 2016 Apr 22. PMID 27209164